CLINICAL TRIAL: NCT01777841
Title: Clinical Pilot:myCare
Brief Title: Mayo Clinic Health Connection Discovery Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, DJCook, Professor, Mayo Medical School, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 11-008757
Record Dates: First submitted 2013-01-24; First posted 2013-01-29 (Estimated); Last update posted 2013-01-29 (Estimated); Status verified 2013-01

CONDITIONS: Surgical Recovery
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electronic Care plan delivery (Other)
  Interventions: Other: Electronic Care plan delivery; Other: Standard care

INTERVENTIONS:
Other: Electronic Care plan delivery
Other: Standard care

SUMMARY:
The MC Health Connection Discovery trial is designed to determine if a new health information system that delviers interactive care plans (delivered by mobile) to patients can impact post-surgical recovery.

ELIGIBILITY:
Inclusion Criteria:

Patients will be English speaking adults without visual or hearing impairments that would prevent use of the Ipad program. Target population will be older than 50 years of age. We will include patients who are undergoing coronary artery bypass grafting, valve repair or replacement or both at St. Mary's Hospital-Rochester, Minnesota. We will also be including family members 18 years of age and over, that may be the primary non-patient user of the iPad.

Exclusion Criteria:

Patients who do not meet inclusion criteria or who are predicted to have very short or very long hospital stays would not be candidates for the program which is designed for a standard 5, 6 or 7 day hospitalization.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2012-02; Primary Completion 2012-11 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Patient usability of IT platform: percent completion of care modules delivered | Day 1 to day 7 of hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Cook DJ, Manning DM, Holland DE, Prinsen SK, Rudzik SD, Roger VL, Deschamps C. Patient engagement and reported outcomes in surgical recovery: effectiveness of an e-health platform. J Am Coll Surg. 2013 Oct;217(4):648-55. doi: 10.1016/j.jamcollsurg.2013.05.003. Epub 2013 Jul 25. PMID 23891066